CLINICAL TRIAL: NCT02685670
Title: A Phase I/II Study of Competitive Transfer of αCD19-TCRz-CD28 and αCD19-TCRz-CD137 Chimeric Antigen Receptor T-Cells in Patients With Refractory CD19+ B-lineage Leukemia/Lymphoma
Brief Title: Competitive Transfer of αCD19-TCRz-CD28 and αCD19-TCRz-CD137 CAR-T Cells for B-cell Leukemia/Lymphoma
Acronym: MatchCART
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Chengzhi, Director of Department of Hematology, The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHHUTCM20160106
Record Dates: First submitted 2016-02-14; First posted 2016-02-19 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Hematopoietic/Lymphoid Cancer; Adult Acute Lymphoblastic Leukemia in Remission; B-cell Adult Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mixed CD19CAR transfer (Experimental): All subjects will be infused with αCD19-TCRz-CD28 and αCD19-TCRz-CD137 CAR-T cells in equal number
  Interventions: Biological: anti-CD19 CAR-T; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: anti-CD19 CAR-T — Ex vivo-expanded autologous T cells modified to express CD19 CAR
Drug: Fludarabine
Drug: Cyclophosphamide

SUMMARY:
This is a single-arm open-label phase I/II study to determine the relative superiority of αCD19-TCRζ-CD28 and αCD19-TCRζ-CD137 CAR-T Cells in safety, efficacy and engraftment potential in patients with CD19+ B-lineage leukemia and lymphoma. Recently, cancer immunotherapy, treatments aiming to arm patients with immunity specifically against cancer cells, has emerged as a promising therapeutic strategy. Clinical trials utilizing CARs against B cell malignancies have demonstrated remarkable potential. In this trial, all subjects will be competitively infused with αCD19-TCRz-CD28 and αCD19-TCRz-CD137 CAR-T cells in equal number to test a hypothesis that CD137-costimulation can promote the persistence and engraftment of CAR-T cells and this superiority can lead to improved progression-free survival.

DETAILED DESCRIPTION:
Primary objectives

1. To determine the safety and feasibility of adoptive transfer of T cells modified to express CD19-specific chimeric antigen receptor (CD19CAR) for treatment of leukemia and lymphoma

Secondary objectives

1. To measure the efficacy of anti-tumor responses after CD19CAR T cell infusion
2. To determine if CD19CAR T cells engineered with 4-1BB signaling domain is superior to that with CD28 signaling domain for their homing and persistence after CD19CAR T cell infusion

ELIGIBILITY:
Inclusion Criteria:

1. 5 Years to 70 Years, Male and female;
2. Expected survival > 12 weeks;
3. Performance score 0-2;
4. Histologically confirmed as CD19-positive lymphoma/leukemia and who meet one of the following conditions;

   * Patient receive at least 2-4 prior combination chemotherapy regimens (not including single agent monoclonal antibody therapy) and fail to achieve CR; or have disease recurrence; or not eligible for allogeneic stem cell transplantation; or disease responding or stable after most recent therapy but refused further treatment;
   * Disease recurrence after stem cell transplantation;
   * Diagnosis as lymphoma, but refuse conventional treatment such as chemotherapy, radiation, stem cell transplantation and monoclonal antibody therapy
5. Creatinine < 2.5 mg/dl;
6. ALT/AST < 3x normal;
7. Bilirubin < 2.0 mg/dl;
8. Adequate venous access for apheresis, and no other contraindications for leukapheresis;
9. Take contraceptive measures before recruit to this trial;
10. Written voluntary informed consent is given.

Exclusion Criteria:

1. Patients with symptoms of central nervous system
2. Accompanied by other malignant tumor
3. Active hepatitis B or C, HIV infection
4. Any other diseases could affect the outcome of this trial
5. Suffering severe cardiovascular or respiratory disease
6. Poorly controlled hypertension
7. A history of mental illness and poorly controlled
8. Taking immunosuppressive agents within 1 week due to organ transplantation or other disease which need long-lasting administration
9. Occurrence of unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolic events 30 days prior to assignment
10. Reaching a steady dose if receiving anticoagulant therapy before assignment
11. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
12. Pregnant or lactating women
13. Subject suffering disease affects the understanding of informed consent or comply with study protocol.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Safety (incidence of adverse events defined as dose-limited toxicity) | 30 days

SECONDARY OUTCOMES:
Overall complete remission rate | 8 weeks
Survival of CAR T cells in circulation measured by flow cytometry and PCR | 1 year
Duration of remission | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Cheng, M.D., Principal Investigator — The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- Henan Province of TCM, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided